CLINICAL TRIAL: NCT00073736
Title: A Phase 1/2 Open-Label Study to Assess the Safety, Tolerability, and Pharmacokinetics of Intravenous Infusion of MB07133 in Subjects With Unresectable Hepatocellular Carcinoma and Child-Pugh Class A Liver Function
Brief Title: Safety and Tolerability of I.V. Infusion of MB07133 in Patients With Unresectable Hepatocellular Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ligand Pharmaceuticals (Industry)
Responsible Party: Director, Project Management, Ligand Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC-101
Record Dates: First submitted 2003-12-03; First posted 2003-12-05 (Estimated); Last update posted 2011-08-12 (Estimated); Status verified 2011-08

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular; Carcinoma; Liver; Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Carcinoma; Neoplasms | interventions — 4-amino-1-(5-O-(2-oxo-4-(4-pyridyl)-1,3,2-dioxaphosphorinan-2-yl)arabinofuranosyl)-2(1H)-pyrimidinone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- MB07133 Dose Level 1 (Experimental): 7-day continuous infusion in 28-day cycles
  Interventions: Drug: MB07133 300mg/m2/day
- MB07133 Dose Level 2 (Experimental): 7-day continuous infusion in 28-day cycles
  Interventions: Drug: MB07133 600 mg/m2/day
- MB07133 Dose Level 3 (Experimental): 7-day continuous infusion in 28-day cycles
  Interventions: Drug: MB07133 1200 mg/m2/day
- MB07133 Dose Level 4 (Experimental): 7-day continuous infusion in 28-day cycles
  Interventions: Drug: MB07133 1800 mg/m2/day
- MB07133 Dose Level 5 (Experimental): 7-day continuous infusion in 28-day cycles
  Interventions: Drug: MB07133 2400 mg/m2/day

INTERVENTIONS:
Drug: MB07133 300mg/m2/day — 7-day continuous infusion in 28-day cycles
  Arms: MB07133 Dose Level 1
Drug: MB07133 600 mg/m2/day — 7-day continuous infusion in 28-day cycles
  Arms: MB07133 Dose Level 2
Drug: MB07133 1200 mg/m2/day — 7-day continuous infusion in 28-day cycles
  Arms: MB07133 Dose Level 3
Drug: MB07133 1800 mg/m2/day — 7-day continuous infusion in 28-day cycles
  Arms: MB07133 Dose Level 4
Drug: MB07133 2400 mg/m2/day — 7-day continuous infusion in 28-day cycles
  Arms: MB07133 Dose Level 5

SUMMARY:
Hepatocellular carcinoma (HCC) is the most common primary cancer of the liver. MB07133 is being developed for the treatment of inoperable HCC, using a platform technology known as HepDirectTM, which enables drugs to be targeted specifically to the liver. The objective for this study is to determine the safety and tolerability of MB07133.

DETAILED DESCRIPTION:
To determine the maximum tolerated dose of MB07133 when administered as a 7-day continuous i.v. To characterize the safety profile and the pharmacokinetics of MB07133 and metabolites during and after continuous infusion. To determine the effect of MB07133 on hepatocellular carcinoma (HCC) tumor size.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of local unresectable HCC confirmed by histology using fine needle aspirate (FNA) or liver biopsy. "Local" is defined as disease either restricted to the liver or contiguous with the liver and no identifiable extrahepatic disease.
* Patients with Child-Pugh Class A liver function. For purposes of this trial, an eligible patient must not have Encephalopathy or Ascites and the total Child-Pugh score cannot be greater than 6 at baseline
* Males or females 18 years of age or older
* Ability to provide written informed consent before initiation of any study-related procedures and ability, in the opinion of the Principal Investigator, to comply with all the requirements of the study
* Male and female subjects who are surgically sterile, who remain abstinent, or who agree to practice double barrier forms of birth control from screening through 30 days (females) and 90 days (males), from the last dose of study medication

Exclusion Criteria:

* History of or presence of clinically significant acute or unstable cardiovascular, cerebrovascular (stroke), renal, GI, pulmonary, immunological (with the exception of the presence of hepatitis B virus [HBV], HCV hepatitis, or cirrhosis), endocrine, or central nervous system disorders
* Patient has a history of cancer other than hepatocellular (excluding resected basal cell carcinoma; or curatively resected stage 1 or less cervical cancer if disease free for 5 years or more).
* Patients with distant metastasis or extrahepatic disease
* An Eastern Cooperative Oncology Group (ECOG) performance status score of greater than or equal to 2
* Current encephalopathy or current treatment for encephalopathy
* History of drug or alcohol abuse within 6 months before screening
* History of, or current clinically significant mental disorder or an antagonistic personality that compromises the validity of the informed consent
* A documented variceal hemorrhage within 4 months of screening
* Neutrophil count less than or equal to 1,500/mm3, platelet count less than or equal to 100,000/mm3, hemoglobin less than or equal to 8.5 g/dL, or a Prothrombin Time (INR) greater than 1.3 (vitamin K supplementation allowed)
* Serum creatinine greater than 1.1 times the upper limit of normal
* History of human immunodeficiency virus or acquired immune deficiency syndrome
* Use of an investigational drug or product or participation in a drug study within 30 days before dosing
* Liver function defined as: serum bilirubin greater than 1.5 times the upper limit of normal or an aspartate aminotransferase (AST) or alanine aminotransferase (ALT) greater than 5 times upper limit of normal, or serum albumin less than 3.2 g/dL
* History of gout or abnormal uric acid metabolism
* The clinical presence of ascites
* Treatment of HCC within 30 days of screening by chemotherapy or treatment of the target lesion(s) by chemoembolization, PEI, or surgery
* Radiofrequency ("RF") ablation of the target lesion(s) within 60 days of screening
* Subjects with a life expectancy of less than 12 weeks
* Subjects having received an organ transplant
* Subjects currently receiving coumadin or heparin
* Pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2003-09; Primary Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 7-day continuous infusion every 28-days as tolerated
  To determine the dose-limiting toxicities (DLT) of MB07133; To determine the maximum-tolerated continuous infusion dose (MTD) of MB07133

SECONDARY OUTCOMES:
Determine effect of MB07133 on tumor size | 28 day cycles
  To determine the effect on HCC tumor size by using CT scanning, alpha-fetoprotein (AFP) concentration, and performance status.

CONTACTS AND LOCATIONS:
Overall Officials: Isabela Niculae, MPH, Study Director — Metabasis Therapeutics, Inc.
Locations (4):
- University of California at Irvine, Orange, California, United States
- Prince of Wales Hospital - Comprehensive Cancer Trial Unit, Shatin, New Territories, Hong Kong
- Taiwan (2):
  - Tri-Services General Hospital, Taipei, Nei Hu District
  - Chang-Gung Memorial Hospital, Taipei, Taoyuan County